CLINICAL TRIAL: NCT03249168
Title: Preoperative Duloxetine to Prevent Postoperative Shoulder Pain After Gynecological Laparoscopies
Brief Title: Duloxetine for Post Laparoscopic Shoulder Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mina fayez ghalyoom, principal invstigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MFGA
Record Dates: First submitted 2017-07-21; First posted 2017-08-15 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Post Laparoscopic Shoulder Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Experimental): Duloxetine 60mg orally 12 hours before surgery
  Interventions: Drug: Duloxetine 60mg
- Control group (Active Comparator): Placebo (glucose powder in a tablet) orally 12 hours before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine 60mg — tablet
  Arms: case group
Drug: Placebo — Tablet
  Arms: Control group

SUMMARY:
Despite recent advances in minimal invasive surgery, postoperative pain control remains a challenge for both surgeons and anesthesiologists . Currently, laparoscopy has an obvious favor for both diagnostic and therapeutic procedures of pelvic and abdomen; while it is minimally invasive, has less pain, and needs less postoperative analgesic use compared with open surgeries . Shoulder pain is a frequent problem following laparoscopic procedure

DETAILED DESCRIPTION:
Many patients may feel much more discomfort from their shoulder pain than incision pain . Post laparoscopic shoulder pain is caused by irritation and/or injury of the diaphragm and phrenic nerve by local acidosis and irritative effect of carbon dioxide during pneumoperitoneum or distention forces on the diaphragm. Duloxetine is a selective serotonin and norepinephrine reuptake inhibitor antidepressant . It is used to treat major depressive disorder in adults. Duloxetine is also used to treat general anxiety disorder. It is also used in adults to treat fibromyalgia (a chronic pain disorder), or chronic muscle or joint pain (such as low back pain and osteoarthritis pain). Duloxetine is also used to treat diabetic neuropathy. Previous studies focused on the use of gabapentin and pregabalin (both are antineuropathic pain medications) to prevent post laparoscopic shoulder pain after laparoscopic ovarian cystectomy and laparoscopic cholecystectomy showed favorable results and since duloxetine is an antineuropathic pain medications we assume its use will ameliorate diaphragmatic irritation and hencepost laparoscopic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females
* Patient consent
* Patients with ASA class I-II
* Elective gynecological laparoscopy

Exclusion Criteria:

* Body Mass Index ≥ 40
* Consuming any pain killers routinely within 48 hours before the surgery
* Smoking, drug abuse
* Patients with major psychiatric disorders, epilepsy or history of convulsion
* Any known kidney or hepatic disorders
* History of any other pervious laparotomy, laparoscopy, or other pelvic manipulation or pathology except normal vaginal delivery
* History of chest or mediastinal surgery or pathology
* Recent flu (six weeks before surgery)
* Suspected to malignancy as pathology
* Those who complained from shoulder pain just before surgery in the first Visual Analog Scale assessment.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
post laparoscopic shoulder pain | 12 hours after surgery
  The presence and severity of Post laparoscopic shoulder pain will be recorded using a Visual Analog Scale

SECONDARY OUTCOMES:
sedation | 12 hours after surgery
  Ramsey Sedation Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Valadan M, Banifatemi S, Yousefshahi F. Preoperative Gabapentin to Prevent Postoperative Shoulder Pain After Laparoscopic Ovarian Cystectomy: A Randomized Clinical Trial. Anesth Pain Med. 2015 Dec 5;5(6):e31524. doi: 10.5812/aapm.31524. eCollection 2015 Dec. PMID 26705527
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pubmed/26705527